CLINICAL TRIAL: NCT00911053
Title: Melatonin for Circadian Sleep Disorders in the Blind
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unique provision in the American Recovery and Reinvestment Act prevented approval of second year no-cost-extension in which completion of analyses were planned.
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: R01EY018312 (NIH); NCT00686907 (obsolete NCT alias)
Record Dates: First submitted 2009-05-07; First posted 2009-06-01 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Insomnia; Blindness; Daytime Sleepiness
Keywords: melatonin; sleep; blindness; blind individuals
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Blindness; Disorders of Excessive Somnolence | interventions — Melatonin; Light

STUDY DESIGN:
Who Masked: Participant

ARMS (5):
- Baseline (No Intervention)
- Melatonin (Experimental): Subjects will be administered melatonin.
  Interventions: Drug: Melatonin
- Light (Experimental)
  Interventions: Behavioral: Light
- Regular Sleep Schedule (Experimental)
  Interventions: Behavioral: Regular Sleep Schedule
- Longitudinal Monitoring (No Intervention): Optional longitudinal study, an extension of the first study stage, for subjects whose rhythms are not clearly free-running.

INTERVENTIONS:
Drug: Melatonin — Melatonin will be administered under FDA IND #26,318, doses between 0.025 mg and 20 mg.
  Arms: Melatonin
Behavioral: Regular Sleep Schedule — Subjects will maintain a regular sleep schedule of their choosing.
  Arms: Regular Sleep Schedule
Behavioral: Light — Subjects will be exposed to light.
  Arms: Light

SUMMARY:
This research project consists of a three part study with five embedded sub studies. The first study phase identifies "body rhythms" of sleepiness/wakefulness and of melatonin levels for each subject (including sub-study 1). The second study phase identifies the optimum dose and timing of melatonin for regulating each individual's 24-hour sleep/waking cycle (including sub-study 2). The third study phase introduces a new independent variable, light (including sub-studies 3 and 4). Sub-study 5 is an optional longitudinal study.

Sub-study 1 looks at how keeping a regular sleep schedule affects the body's natural rhythm. Sub-study 2 looks at how individuals metabolize melatonin. Sub-study 3 tests how individuals' endogenous melatonin production responds to bright outdoor light and Sub-study 4 tests a previous finding that artificial bright light exposed daily behind the knee can regulate the body clock. Sub-study 5 is an optional longitudinal study, an extension of the first study stage, for subjects whose rhythms are not clearly free-running.

ELIGIBILITY:
Inclusion criteria:

* blindness for at least one year, verified by an ophthalmologic exam
* ability to comply with the requirements of the experimental protocol
* competency to sign informed consent

Exclusion criteria (as determined by medical history and/or physical examination):

* abnormal heart, liver or kidney function
* a current Axis I psychiatric or substance abuse disorder according to the DSM-IV Manual
* possibly external demands that limit the ability to maintain a regular schedule (e.g., night shift work)
* sexually active female subjects of child-bearing potential will be asked to avoid pregnancy using accepted methods and will be notified that the effects of melatonin on a fetus are not known (we will ask subjects monthly if they are pregnant or trying to become pregnant)
* if a subject reports she is pregnant or is trying to become pregnant anytime during her study participation, any study medications (melatonin or placebo) will be immediately withdrawn and the subject will be excluded from the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 1997-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Lewy, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Period: Overall Study
Arm/Group | Baseline | Melatonin | Light | Regular Sleep Schedule | Longitudinal Monitoring
Started | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Baseline | Melatonin | Light | Regular Sleep Schedule | Longitudinal Monitoring | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Treatment Effects on Circadian Phase Will be Assessed During Each Trial by Measuring the Timing of Endogenous Melatonin Secretion.
Time Frame: 1 year
Population: as for baseline characteristics
Arm/Group | Baseline | Melatonin | Light | Regular Sleep Schedule | Longitudinal Monitoring
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Treatment Effects on Sleep and Alertness Will be Assessed by Daily Diaries and Daily Wrist Actigraphic Monitoring. Subjective Benefits Will be Assessed With Daily Ratings of Alertness and Vigor.
Time Frame: 1 year
Population: as for baseline characteristics
Arm/Group | Baseline | Melatonin | Light | Regular Sleep Schedule | Longitudinal Monitoring
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The PI has retired from the institution. Sincere efforts were made to contact the PI/study team members, but were unsuccessful. No study data are available.
Arm/Group | Baseline | Melatonin | Light | Regular Sleep Schedule | Longitudinal Monitoring
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Analyses were not completed because a unique provision in the American Recovery and Reinvestment Act (ARRA) of 2009 funding source unexpectedly prevented approval of a second year no-cost-extension in which completion of analyses were planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No